CLINICAL TRIAL: NCT07290699
Title: INtensive Cholesterol-Lowering With recatIcimab combiNation in Emergency PCI for Acute Myocardial Infarction: A Randomized Controlled Trial
Brief Title: Intensive Cholesterol-Lowering Within 24 Hours of PCI Perioperative Period
Acronym: INCLINE-AMI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: First Affiliated Hospital of Gannan Medical University (Other); Jiujiang No.1 People's Hospital (Other); First People's Hospital of FuZhou (Other); Yueyang Central Hospital (Other); The First People's Hospital of Changde City (Other); ZhuZhou Central Hospital (Other); Xiangtan Central Hospital (Other); Loudi Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-I-2025-098
Record Dates: First submitted 2025-11-16; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation Myocardial Infarction (MI)
Keywords: Acute myocardial infarction; Recaticimab; PCSK9 inhibitor
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intensive lipid-lowering within 24 hours during the perioperative period of AMI (standard treatment + PCSK9 inhibitors)；Recaticimab 450 mg once every 12 weeks
  Interventions: Drug: Recaticimab
- Control group (No Intervention): Standard treatment (antiplatelet drugs, 20mg atorvastatin / 10mg rosuvastatin ± cholesterol absorption inhibitors)

INTERVENTIONS:
Drug: Recaticimab — Recaticimab 450 mg once every 12 weeks. Group 1 (G1, experimental group): Intensive lipid-lowering therapy within 24 hours during the perioperative period of AMI (standard treatment + PCSK9 inhibitors), treatment for 6 months; Group 2 (G2, control group): standard treatment (antiplatelet drugs, 20 mg atorvastatin/10 mg rosuvastatin ± cholesterol absorption inhibitors). After 6 months, both groups continued with guideline-recommended conventional treatment.
  Arms: Intervention Group

SUMMARY:
This project team is conducting a multicenter randomized controlled study, aiming to administer PCSK9 inhibitors subcutaneously as early as possible within 24 hours during the perioperative period of AMI (included <24h STEMI and NSTEMI), and subsequently once every 12 weeks for a total of 6 months, followed by step-down therapy according to guideline-recommended lipid-lowering strategies based on LDL-C target levels. The study will evaluate changes in blood lipids and inflammatory markers during hospitalization and at follow-up visits at 1, 3, 6, 9, and 12 months, as well as the incidence of MACE events. Safety will also be assessed, including liver enzymes, kidney function, and other adverse reactions. Compared with conventional treatment, the study will test efficacy and ultimately clarify that early combined use of PCSK9 inhibitors during the perioperative period of AMI patients can safely and effectively reduce LDL-C, control systemic inflammatory responses, and improve the incidence of MACE events.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized controlled trial, with the Second Affiliated Hospital of Nanchang University as the leading center and 80 sub-centers established. The enrollment period is from September 1, 2025, to August 30, 2027, with a follow-up of 1 year. A total of 2,442 patients who meet the inclusion criteria will be randomly assigned to: Group 1 (G1, experimental group): intensive lipid-lowering therapy within 24 hours during the perioperative period of AMI (standard treatment + PCSK9 inhibitors) for 6 months; Group 2 (G2, control group): standard lipid-lowing treatment (20 mg atorvastatin/10 mg rosuvastatin ± cholesterol absorption inhibitors). After 6 months, both groups will continue treatment according to guideline-recommended standard therapy.

Randomization method: All eligible patients entering the respective groups will be randomly obtained a random number. The maximum follow-up period is 1 year. Safety evaluation includes monitoring all adverse events (AEs), serious adverse events (SAEs), as well as regular monitoring of vital signs and clinical laboratory tests.

Each center will screen hospitalized AMI patients according to inclusion and exclusion criteria. Baseline data will be entered into the CRF form for the first time, including basic patient information, admission details, laboratory and instrument examinations, surgical procedure details, postoperative medications, and occurrence of adverse events during hospitalization. After discharge, follow-up visits will be conducted at 1 month, 3 months, 6 months, 9 months, and 1 year, inquiring about current health status and medication usage, and recording the occurrence of endpoint events and lipid levels in the follow-up section of the CRF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Meet the definition of acute myocardial infarction according to the "2019 Guidelines for the Diagnosis and Treatment of Acute ST-Segment Elevation Myocardial Infarction", including STEMI and NSTEMI with onset <24 hours;
* Able to understand and voluntarily sign the informed consent form.

Exclusion Criteria:

* Severe mental disorders that prevent the expression of consent;
* Severe heart failure (Killip class III or IV) or cardiogenic shock;
* According to the investigator's judgment, the presence of significant other abnormal signs, laboratory findings, or clinical conditions (such as tumors, shock, liver or kidney failure, etc.) that make participation unsuitable;
* Investigator's judgment that the subject cannot complete long-term follow-up;
* Intolerance to statins or cholesterol absorption inhibitors;
* Intolerance to injections;
* Subjects who received PCSK9 inhibitor treatment or participated in other PCSK9 inhibitor studies within 4 months before randomization;
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2442 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
MACE | From enrollment to the end of treatment at 12 months
  The primary endpoint was 1-year MACE (major adverse cardiovascular and cerebrovascular events, including cardiac death, non fatal myocardial infarction, non fatal stroke, or hospitalization due to unplanned unstable angina and coronary revascularization).

SECONDARY OUTCOMES:
LDL-C reduction absolute value | From enrollment to the end of treatment at 12 months, and record the values for every 1, 3, 6, 9, and 12 months if possible.
  LDL-C reduction absolute value means, it refers to the LDL-C value measured in the 12th month minus the LDL-C value measured at baseline.
LDL-C targets achieved rate | From enrollment to the end of treatment at 12 months, and record the values for every 1, 3, 6, 9, and 12 months if possible
  LDL-C targets achieved rate, it refers to whether the LDL-C at the 12th month has reached the target value recommended by the guidelines for the patient.
Changes in Lp (a) levels | From enrollment to the end of treatment at 12 months, and record the values for every 1, 3, 6, 9, and 12 months if possible
  Changes in Lp (a) levels, it refers to the changes in baseline Lp (a) levels and Lp (a) levels at the 12th month
Changes in the size of carotid plaques | From baseline to the mid at 6 months and end of treatment at the 12 months
  Record changes in carotid plaque size at baseline and 12-month follow-up
Observation indicators of safety | From enrollment to the end of treatment at 1, 3, 6, 9 ,12 months.
  Adverse events (AEs) are defined as any adverse medical events that occur during the period from the signing of informed consent by clinical trial subjects until the completion of the study.
The occurrence rate of MACE events in 6 months | From enrollment to the end of treatment at 6 months.
  6-month incidence of MACE events (referring to cardiac death, non fatal myocardial infarction, hospitalization due to unstable angina, and coronary revascularization);
Cardiac death | From enrollment to the end of treatment at 6 months and 1 year
  Record cardiac death at 6 months and 1 year
Non fatal myocardial infarction | From enrollment to the end of treatment at 6 months and 1 year.
  Recard non fatal myocardial infarction at 6 months and 1 year.
Non fatal stroke | From enrollment to the end of treatment at 6 months and 1 year
  Record non fatal stroke at 6 months and 1 year
Hospitalization due to unplanned unstable angina and coronary revascularization | From enrollment to the end of treatment at 6 months and 1 year.
  Record hospitalization due to unplanned unstable angina and coronary revascularization at 6 months and 1 year.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654
- [Result] Rao SV, O'Donoghue ML, Ruel M, Rab T, Tamis-Holland JE, Alexander JH, Baber U, Baker H, Cohen MG, Cruz-Ruiz M, Davis LL, de Lemos JA, DeWald TA, Elgendy IY, Feldman DN, Goyal A, Isiadinso I, Menon V, Morrow DA, Mukherjee D, Platz E, Promes SB, Sandner S, Sandoval Y, Schunder R, Shah B, Stopyra JP, Talbot AW, Taub PR, Williams MS. 2025 ACC/AHA/ACEP/NAEMSP/SCAI Guideline for the Management of Patients With Acute Coronary Syndromes: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2025 Apr;151(13):e771-e862. doi: 10.1161/CIR.0000000000001309. Epub 2025 Feb 27. PMID 40014670
- [Result] Raber L, Ueki Y, Otsuka T, Losdat S, Haner JD, Lonborg J, Fahrni G, Iglesias JF, van Geuns RJ, Ondracek AS, Radu Juul Jensen MD, Zanchin C, Stortecky S, Spirk D, Siontis GCM, Saleh L, Matter CM, Daemen J, Mach F, Heg D, Windecker S, Engstrom T, Lang IM, Koskinas KC; PACMAN-AMI collaborators. Effect of Alirocumab Added to High-Intensity Statin Therapy on Coronary Atherosclerosis in Patients With Acute Myocardial Infarction: The PACMAN-AMI Randomized Clinical Trial. JAMA. 2022 May 10;327(18):1771-1781. doi: 10.1001/jama.2022.5218. PMID 35368058
- [Result] Koskinas KC, Windecker S, Pedrazzini G, Mueller C, Cook S, Matter CM, Muller O, Haner J, Gencer B, Crljenica C, Amini P, Deckarm O, Iglesias JF, Raber L, Heg D, Mach F. Evolocumab for Early Reduction of LDL Cholesterol Levels in Patients With Acute Coronary Syndromes (EVOPACS). J Am Coll Cardiol. 2019 Nov 19;74(20):2452-2462. doi: 10.1016/j.jacc.2019.08.010. Epub 2019 Aug 31. PMID 31479722
- [Result] Ferri N, Ruscica M, Lupo MG, Vicenzi M, Sirtori CR, Corsini A. Pharmacological rationale for the very early treatment of acute coronary syndrome with monoclonal antibodies anti-PCSK9. Pharmacol Res. 2022 Oct;184:106439. doi: 10.1016/j.phrs.2022.106439. Epub 2022 Sep 12. PMID 36100012
- [Result] Cannon CP, Braunwald E, McCabe CH, Rader DJ, Rouleau JL, Belder R, Joyal SV, Hill KA, Pfeffer MA, Skene AM; Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 Investigators. Intensive versus moderate lipid lowering with statins after acute coronary syndromes. N Engl J Med. 2004 Apr 8;350(15):1495-504. doi: 10.1056/NEJMoa040583. Epub 2004 Mar 8. PMID 15007110
- [Result] Schwartz GG, Olsson AG, Ezekowitz MD, Ganz P, Oliver MF, Waters D, Zeiher A, Chaitman BR, Leslie S, Stern T; Myocardial Ischemia Reduction with Aggressive Cholesterol Lowering (MIRACL) Study Investigators. Effects of atorvastatin on early recurrent ischemic events in acute coronary syndromes: the MIRACL study: a randomized controlled trial. JAMA. 2001 Apr 4;285(13):1711-8. doi: 10.1001/jama.285.13.1711. PMID 11277825
- [Result] Patti G, Pasceri V, Colonna G, Miglionico M, Fischetti D, Sardella G, Montinaro A, Di Sciascio G. Atorvastatin pretreatment improves outcomes in patients with acute coronary syndromes undergoing early percutaneous coronary intervention: results of the ARMYDA-ACS randomized trial. J Am Coll Cardiol. 2007 Mar 27;49(12):1272-8. doi: 10.1016/j.jacc.2007.02.025. PMID 17394957
- [Result] Huang D, Wu H, Zhou J, Zhong X, Gao W, Ma Y, Qian J, Ge J. Intravenous nicorandil during primary percutaneous coronary intervention in patients with ST-Elevation myocardial infarction: Rationale and design of the Clinical Efficacy and Safety of Intravenous Nicorandil (CLEAN) trial. Am Heart J. 2022 Feb;244:86-93. doi: 10.1016/j.ahj.2021.11.005. Epub 2021 Nov 14. PMID 34785173
- [Result] Lopes RD, de Barros E Silva PGM, de Andrade Jesuino I, Santucci EV, Barbosa LM, Damiani LP, Nakagawa Santos RH, Laranjeira LN, Dall Orto FTC, Beraldo de Andrade P, de Castro Bienert IR, Alexander JH, Granger CB, Berwanger O. Timing of Loading Dose of Atorvastatin in Patients Undergoing Percutaneous Coronary Intervention for Acute Coronary Syndromes: Insights From the SECURE-PCI Randomized Clinical Trial. JAMA Cardiol. 2018 Nov 1;3(11):1113-1118. doi: 10.1001/jamacardio.2018.3408. PMID 30264159
- [Result] Wu XD, Ye XY, Liu XY, Lin Y, Lin X, Li YY, Ye BH, Sun JC. Benefits of intensive lipid-lowering therapies in patients with acute coronary syndrome: a systematic review and meta-analysis. Ann Med. 2024 Dec;56(1):2389470. doi: 10.1080/07853890.2024.2389470. Epub 2024 Aug 10. PMID 39126262
- [Result] Gaba P, O'Donoghue ML, Park JG, Wiviott SD, Atar D, Kuder JF, Im K, Murphy SA, De Ferrari GM, Gaciong ZA, Toth K, Gouni-Berthold I, Lopez-Miranda J, Schiele F, Mach F, Flores-Arredondo JH, Lopez JAG, Elliott-Davey M, Wang B, Monsalvo ML, Abbasi S, Giugliano RP, Sabatine MS. Association Between Achieved Low-Density Lipoprotein Cholesterol Levels and Long-Term Cardiovascular and Safety Outcomes: An Analysis of FOURIER-OLE. Circulation. 2023 Apr 18;147(16):1192-1203. doi: 10.1161/CIRCULATIONAHA.122.063399. Epub 2023 Feb 13. PMID 36779348
- [Result] Steg PG, Szarek M, Bhatt DL, Bittner VA, Bregeault MF, Dalby AJ, Diaz R, Edelberg JM, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Lecorps G, Mahaffey KW, Moryusef A, Ostadal P, Parkhomenko A, Pordy R, Roe MT, Tricoci P, Vogel R, White HD, Zeiher AM, Schwartz GG. Effect of Alirocumab on Mortality After Acute Coronary Syndromes. Circulation. 2019 Jul 9;140(2):103-112. doi: 10.1161/CIRCULATIONAHA.118.038840. Epub 2019 May 23. PMID 31117810
- [Result] Sawhney JPS, Mullasari A, Kahali D, Mehta V, Nair T, Kaul U, Hirematth MS. Short- and long-term follow-up of antithrombotic management patterns in patients hospitalized with acute coronary syndrome: Indian subgroup of EPICOR Asia study. Indian Heart J. 2019 Jan-Feb;71(1):25-31. doi: 10.1016/j.ihj.2018.12.005. Epub 2019 Jan 3. PMID 31000179
- [Result] Song J, Murugiah K, Hu S, Gao Y, Li X, Krumholz HM, Zheng X; China PEACE Collabortive Group. Incidence, predictors, and prognostic impact of recurrent acute myocardial infarction in China. Heart. 2020 Sep 16;107(4):313-8. doi: 10.1136/heartjnl-2020-317165. Online ahead of print. PMID 32938773
- [Result] Chi G, Lee JJ, Kazmi SHA, Fitzgerald C, Memar Montazerin S, Kalayci A, Korjian S, Heise M, Deckelbaum LI, Libby P, Bhatt DL, Gibson CM. Early and late recurrent cardiovascular events among high-risk patients with an acute coronary syndrome: Meta-analysis of phase III studies and implications on trial design. Clin Cardiol. 2022 Mar;45(3):299-307. doi: 10.1002/clc.23773. Epub 2022 Jan 12. PMID 35019162
- [Result] Cholesterol Treatment Trialists' (CTT) Collaboration; Baigent C, Blackwell L, Emberson J, Holland LE, Reith C, Bhala N, Peto R, Barnes EH, Keech A, Simes J, Collins R. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet. 2010 Nov 13;376(9753):1670-81. doi: 10.1016/S0140-6736(10)61350-5. Epub 2010 Nov 8. PMID 21067804
- [Result] Gargiulo P, Basile C, Galasso G, Bellino M, D'Elia D, Patti G, Bosco M, Prinetti M, Ando G, Campanella F, Taverna G, Calabro P, Cesaro A, Fimiani F, Catalano A, Varbella F, Corleto A, Barilla F, Muscoli S, Musumeci G, Delnevo F, Giallauria F, Napoli R, Porto I, Polimeni A, Quarta R, Maloberti A, Merlini PA, De Luca L, Casu G, Brunetti ND, Crisci M, Paloscia L, Bilato C, Indolfi C, Marzano F, Fontanarosa S, Buonocore D, Parlati ALM, Nardi E, Prastaro M, Soricelli A, Salvatore M, Paolillo S, Perrone-Filardi P, Cuomo G, Testa C, Passaretti G, Vallefuoco G, Romano A, Dell'Anno R, Merolla A, Iannone FP. Strike early-strike strong lipid-lowering strategy with proprotein convertase subtilisin/kexin type 9 inhibitors in acute coronary syndrome patients: real-world evidence from the AT-TARGET-IT registry. Eur J Prev Cardiol. 2024 Nov 11;31(15):1806-1816. doi: 10.1093/eurjpc/zwae170. PMID 38788773
- [Result] Yifan D, Yue M, Yubin Z, Jiapei G, Xun S, Shenghu H, Li Z, Jing Z. The impact of early in-hospital use of PCSK9 inhibitors on cardiovascular outcomes in acute coronary syndrome patients: A systematic review and meta-analysis. Int J Cardiol. 2024 Mar 15;399:131775. doi: 10.1016/j.ijcard.2024.131775. Epub 2024 Jan 9. PMID 38211676